| 1 |
|---|
| 1 |
| 1 |

| Official Title: | Urban Zen Integrative Therapy for Person with |
|-----------------|-----------------------------------------------|
| | Pulmonary Hypertension |
| NCT Number: | NCT03194438 |
| Document Name: | Informed Consent Form |
| Document Date: | April 25, 2017 |

2

3

4

5

# The Ohio State University Combined Consent to Participate in Research and HIPAA Research Authorization

7 8

Feasibility and Acceptability of Integrative Therapy in Symptom Management for Persons with Pulmonary

**Study Title:** 

Hypertension

**Principal Investigator:** 

Mary Elizabeth Happ, Ph.D., RN, FGSA, FAAN

**Sponsor:** 

The Ohio State University College of Nursing

9 10

11

12

13

14

15

16

17

18

19

20

21

22

23

24

25

26

- This is a consent form for research participation. It contains important information about this study and what to expect if you decide to participate. Please consider the information carefully. Feel free to discuss the study with your friends and family and to ask questions before making your decision whether or not to participate.
- Your participation is voluntary. You may refuse to participate in this study. If you decide to take part in the study, you may leave the study at any time. No matter what decision you make, there will be no penalty to you and you will not lose any of your usual benefits. Your decision will not affect your future relationship with The Ohio State University. If you are a student or employee at Ohio State, your decision will not affect your grades or employment status.
- You may or may not benefit as a result of participating in this study. Also, as explained below, your participation may result in unintended or harmful effects for you that may be minor or may be serious depending on the nature of the research.
- You will be provided with any new information that develops during the study that may affect your decision whether or not to continue to participate. If you decide to participate, you will be asked to sign this form and will receive a copy of the form. You are being asked to consider participating in this study for the reasons explained below.

272829

30

31

32

# 1. Why is this study being done?

This study is being done to evaluate if a type of integrative therapy called Urban Zen Integrative Therapy (UZIT) is feasible and acceptable for patients with Pulmonary Hypertension. We also would like to observe what impact this therapy may have for patients dealing with a chronic condition such as Pulmonary Hypertension.

333435

# 2. How many people will take part in this study?

Twenty patients will be asked to take part in this study.

3637

# 3. What will happen if I take part in this study?

 If you agree to take part in this study, you will receive six, individual, weekly sessions of UZIT which will be videotaped. Some of the video recordings will be reviewed to make sure that each UZIT session is provided in a consistent manner throughout the study. After most UZIT sessions, we will ask you to describe about how the session went (semi-structured interview). You will complete questionnaires about your symptoms, activity level, and your quality of life. You will also complete a home practice diary to record how and how long you practice UZIT at home.

UZIT will include the use of 3 essential oils (lavender, lemon, or peppermint), and gentle body movement. It also includes restorative pose which includes light twists, seated forward folds and gentle backward bends. There will also be body-awareness meditation (guided meditation) and energy healing therapy (therapeutic touch). UZIT is a free service and currently available for hospitalized patients at the Ohio State University Wexner Medical Center.

Before each scheduled UZIT study visit, a research staff will remind you of your appointment through a phone call or a text message. We will call/ text you through the preferred method of contact as indicated by you.

### 4. How long will I be in the study?

If you choose to participate, you will be in the study for the period of 6-8 weeks. Each study session will last about 60-90 minutes. Home diary completion will take about 5-10 minutes per week.

#### 5. Can I stop being in the study?

You may leave the study at any time. If you decide to stop participating in the study, there will be no penalty to you, and you will not lose any benefits to which you are otherwise entitled. Your decision will not affect your future relationship with The Ohio State University.

#### 6. What risks, side effects or discomforts can I expect from being in the study?

There is a potential risk of allergic reaction to inhalation of essential oil during the UZIT session, but is considered to be rare. We will take this precaution by having you smell a very small amount of each oil while sitting quietly before you are enrolled in the study.

Some changes in your blood pressure and heart rate related to position change during UZIT practice may occur. Since UZIT is not an exercise program, but rather a mind-body practice with gradual body position change, this risk is small.

When answering survey questions about symptoms or feelings, there is also a potential risk of emotional distress.

There is a small risk of confidentiality breach. We will follow the Institutional Review Board (IRB) guidelines in protecting your privacy pertaining to electronic, hard copy data collection as well as video recording of the sessions.

848586

87

88

82

83

# 7. What benefits can I expect from being in the study?

There may be no direct benefit to you from being in the study. However, possible benefit may include relaxation and/or symptom relief.

89 90

### 8. What other choices do I have if I do not take part in the study?

91 92 93

You may choose not to participate without penalty or loss of benefits to which you are otherwise entitled.

94 95 96

# 9. What are the costs of taking part in this study?

97 98

99

There is no additional costs to you in taking part in this study. UZIT session will be provided to you free of charge. You do not have to pay for parking to attend the UZIT session.

100101

### 10. Will I be paid for taking part in this study?

102103104

Study participants will be paid in the form of \$5.00 grocery store gift cards at the end of each UZIT session. The total amount for the entire study is \$30.00.

105106107

#### 11. What happens if I am injured because I took part in this study?

108109

If you suffer an injury from participating in this study, you should notify the researcher immediately, who will determine if you should obtain medical treatment at The Ohio State University Wexner Medical Center.

111112113

114

110

The cost for this treatment will be billed to you or your medical or hospital insurance. The Ohio State University has no funds set aside for the payment of health care expenses for this study.

115116117

#### 12. What are my rights if I take part in this study?

118119

If you choose to participate in the study, you may discontinue participation at any time without penalty or loss of benefits. By signing this form, you do not give up any personal legal rights you may have as a participant in this study.

121122123

124

125

120

You will be provided with any new information that develops during the course of the research that may affect your decision whether or not to continue participation in the study.

| 1 | 26 |
|---|----|
| 1 | 27 |

You may refuse to participate in this study without penalty or loss of benefits to which you are otherwise entitled.

128129130

131

132

An Institutional Review Board responsible for Human Subjects research at The Ohio State University reviewed this research project and found it to be acceptable, according to applicable state and federal regulations and University policies designed to protect the rights and welfare of participants in research.

133134

135136

137

#### 4.0

# 13. Will my study-related information be kept confidential?

138139140

141

Every effort will be made to keep your study-related information confidential. However, there may be circumstances where this information must be released. For example, personal information regarding your participation in this study may be disclosed if required by state law.

142143144

Also, your records may be reviewed by the following groups (as applicable to the research):

145 146

• Office for Human Research Protections or other federal, state, or international regulatory agencies;

147148

• U.S. Food and Drug Administration;

149 150  The Ohio State University Institutional Review Board or Office of Responsible Research Practices;

151 152 The sponsor supporting the study, their agents or study monitors; and
Your insurance company (if charges are billed to insurance).

153

154 155

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search the website at any time.

157158159

156

# 14. HIPAA AUTHORIZATION TO USE AND DISCLOSE INFORMATION FOR RESEARCH PURPOSES

160161162

# I. What information may be used and given to others?

163

• Past and present medical records;

164

• Research records;

165 166

• Records about phone calls made as part of this research;

167

• Records about your study visits;

168 169 • Information that includes personal identifiers, such as your name, or a number associated with you as an individual;

| 170 | • Information gathered for this research about: |
|---|---|
| 171 | Cardiac Catheterization result |
| 172 | Pulmonary Hypertension medications and other medications |
| 173 | Video- recording of UZIT sessions |
| 174 | Diaries and questionnaires |
| 175 | The diagnosis and treatment of a mental health condition |
| 176 | Hospitalization encounters |
| 177 | II. Who may use and give out information about you? |
| 178 | |
| 179<br>180 | Researchers and study staff. |
| 181<br>182 | III. Who might get this information? |
| 183 | Authorized Ohio State University staff not involved in the study may be aware that |
| 184 | you are participating in a research study and have access to your information; |
| 185<br>186 | • If this study is related to your medical care, your study-related information may be placed in your permanent hospital, clinic or physician's office record; |
| 187 | <ul> <li>Others: The Dissertation committee members who collaborate in this project,</li> </ul> |
| 188 | healthcare providers who manage your care, data safety monitoring board that |
| 189 | review safety data. |
| 190 | 10 view surery data. |
| 191 | IV. Your information may be given to: |
| 192 | <del></del> |
| 193<br>194 | • The U.S. Food and Drug Administration (FDA), Department of Health and Human Services (DHHS) agencies, and other federal and state entities; |
| | · · · · · |
| 195 | • Governmental agencies in other countries; |
| 196<br>197 | <ul> <li>Governmental agencies to whom certain diseases (reportable diseases) must be<br/>reported; and</li> </ul> |
| 198 | <ul> <li>The Ohio State University units involved in managing and approving the research</li> </ul> |
| 199 | study including the Office of Research and the Office of Responsible Research |
| 200 | Practices. |
| 201 | |
| 202 | V. Why will this information be used and/or given to others? |
| 203 | |
| 204 | • To do the research; |
| 205 | To study the results; and |
| 206 | To make sure that the research was done right. |
| 207 | To make out a man are recomment in the mone right. |
| 208 | VI. When will my permission end? |
| 209 | |
| 210 | There is no specified date at which your permission ends unless you withdraw consent. |
| 211 | Your information will be used indefinitely. This is because the information used and |
| 212 | created during the study may be analyzed for many years, and it is not possible to know |
| 213 | when this will be complete. |

| 2 | 1 | 4 |
|---|---|---|

215

216

217 218

> 219 220 221

222 223

224 225

226 227

228

229

230 231

232 233

234

235 236

> 237 238

239 240

241 242

243 244

245 246

247 248

250 251

249

252 253

254

255

256

For questions about your rights as a participant in this study or to discuss other study-

authorization, please contact

related concerns or complaints with someone who is not part of the research team, you

W. Tenth Avenue, Columbus OH 43210 Tel: 614-293-4477.

VII. May I withdraw or revoke (cancel) my permission?

been gathered may still be used and given to others.

X. May I review or copy my information?

related information until the study is completed.

15. Who can answer my questions about the study?

harmed as a result of study participation, you may contact

information?

receive care.

Yes. Your authorization will be good for the time period indicated above unless you

change your mind and revoke it in writing. You may withdraw or take away your

be able to stay in this study. When you withdraw your permission, no new health

permission to use and disclose your health information at any time. You do this by

sending written notice to the researchers. If you withdraw your permission, you will not

information identifying you will be gathered after that date. Information that has already

VIII. What if I decide not to give permission to use and give out my health

treatment. However, if you are being treated as a patient here, you will still be able to

Then you will not be able to be in this research study and receive research-related

IX. Is my health information protected after it has been given to others?

information that is shared may no longer be protected by federal privacy rules.

There is a risk that your information will be given to others without your permission. Any

Signing this authorization also means that you may not be able to see or copy your study-

For questions, concerns, or complaints about the study, or if you feel you have been

For questions related to your privacy rights under HIPAA or related to this research

43210 USA. Phone: 1-614-292-8336 Fax: 1-614-292-7976 Email: Happ.3@osu.edu.

Dr. Mary Beth Happ, Ohio State University College of Nursing, 1585 Neil Ave., Columbus, OH

HIPAA Privacy Manager, the Ohio State University Medical Center, 140 Doan Hall, 410

Page 7 of 9

# CONSENT & AUTHORIZATION

#### IRB Protocol Number: IRB Approval date: Version:

| 257 | may contact Ms. Sandra Meadows in the Office of Responsible Research Practices at 1- |
|---|---|
| 258 | 800-678-6251. |
| 259 | |
| 260 | If you are injured as a result of participating in this study or for questions about a study- |
| 261 | related injury, you may contact |
| 262 | |
| 263 | Dr. Mary Beth Happ, Ohio State University College of Nursing, 1585 Neil Ave., Columbus, OH |
| 264 | 43210 USA. Phone: 1-614-292-8336 Fax: 1-614-292-7976 Email: Happ.3@osu.edu. |
| 265 | |
| 266 | |
| 267 | |

| Signing the consent form | | |
|---|---|---|
| I have read (or someone has read to me) this for participate in a research study. I have had the or answered to my satisfaction. I voluntarily agree | pportunity to ask questions and ha | |
| I am not giving up any legal rights by signing the combined consent and HIPAA research authorized | | `this |
| Printed name of subject | Signature of subject | |
| | Date and time | AM/P |
| Printed name of person authorized to consent for subject (when applicable) | Signature of person authorized to consent (when applicable) | t for subject |
| Relationship to the subject | | AM/P |
| signature(s) above. There are no blanks in this to the participant or his/her representative. | accument. If copy of this form ha | |
| Printed name of person obtaining consent | Signature of person obtaining consent | |
| Printed name of person obtaining consent | Signature of person obtaining consent Date and time | AM/P |
| Witness(es) - May be left blank if not require | Date and time | |
| | Date and time | |
| Witness(es) - May be left blank if not requir | Date and time red by the IRB | |
| Witness(es) - May be left blank if not requir | Date and time red by the IRB Signature of witness | AM/P |
| Witness(es) - May be left blank if not requirements Printed name of witness | Date and time red by the IRB Signature of witness Date and time | AM/I |